CLINICAL TRIAL: NCT03704415
Title: Aggravated Airway Inflammation: Research on Genomics and Optimal Operative Treatment (AirGOs Operative)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Paula Virkkula, Chief Physician in Rhinology, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AirGOs Operative
Record Dates: First submitted 2018-10-08; First posted 2018-10-12 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Sinusitis, Chronic; Asthma; Nasal Polyps; Aspirin Sensitivity
MeSH Terms: conditions — Sinusitis; Bronchiolitis Obliterans Syndrome; Asthma; Nasal Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended (Active Comparator): Extended sinus surgery including all sinuses
  Interventions: Procedure: Extended endoscopic sinus surgery
- Limited (Active Comparator): Limited sinus surgery with partial ethmoidectomy
  Interventions: Procedure: Limited endoscopic sinus surgery

INTERVENTIONS:
Procedure: Extended endoscopic sinus surgery — ESS of all sinuses
  Arms: Extended
Procedure: Limited endoscopic sinus surgery — Partial ethmoidectomy
  Arms: Limited

SUMMARY:
This randomized study compares operative techniques in chronic rhinosinusitis with polyposis (CRSwNP) surgery. It aims to evaluate outcomes in asthma and CRSwNP, safety and costs. The investigators want to see if patients with certain clinical and/or genetic predispositions will benefit from extended surgery. They also aim to find biomarkers for detection and management models for of severe airway inflammation and to further develop markers for progressive disease forms.

DETAILED DESCRIPTION:
Please see study protocol

ELIGIBILITY:
Inclusion Criteria:

* Patient not responding to conservative treatment of 3 months of nasal steroid drops
* Nasal polyp score ≥ 4/8
* SNOT-22 ≥ 30
* Lund-Mackay CT score ≥ 14
* One previous endoscopic sinus surgery or at least one peroral corticosteroid course or at least 3 courses of antibiotics within 2 years

Exclusion Criteria:

* Age <18 years, age > 65 years
* Complication of CRS (f.e. mucocele, invasive fungal rhinosinusitis)
* Other diagnosis than CRSwNP (inverted papilloma, antrochoanal polyp etc.)
* Previous external sinus surgery or Draf 3 procedure (or indication for external approaches or Draf 3
* Bleeding diathesis
* Pregnancy/ breastfeeding
* Cystic fibrosis
* Primary ciliary dyskinesia (PCD)
* Sarcoidosis
* Granulomatosis with polyangitis (GPA)
* Eosinophilic granulomatosis with polyangitis (EGPA)
* Immunosupression (diagnosed Spesific Antibody Deficiency (SAD), common variable immunodeficiency (CVI), HIV or use of biologicals/immunosuppressive medication)
* Immunotherapy
* Daily use of systemic corticosteroids
* Communication problems (f.e. neurological/psychiatric disease, language skills)
* Unlikely to comply
* Other severe disease
* Inability to be operated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Sino-nasal outcome test (SNOT-22) | Baseline, Post-intervention every 3 months during 2 years
  Change from baseline in patient symptoms as measured by the Sino-Nasal Outcomes Test (SNOT-22) survey. Scores are measured from 0-5 in a 22 item validated survey. Total scores range from 0-110 with higher scores indicating greater burden of sinonasal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Virkkula, Docent, Principal Investigator — Helsinki University Central Hospital
Locations (3):
- Finland (2):
  - Department of Otorhinolaryngology, Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices) can be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years after article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT03704415/Prot_SAP_000.pdf